CLINICAL TRIAL: NCT03754504
Title: Evaluation of the Effect of Cranberry Whole Fruit Powder on Gut Microbiota Diversity, Intestinal Health and Metabolic Syndrome in Overweight Individuals: a Proof-of-concept Study
Brief Title: Effects of Cranberry Powder Supplements on Gut Microbiota Diversity and Metabolic Syndrome
Acronym: MICA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laval University (Other)
Collaborators: Naturex (Other)
Responsible Party: Principal Investigator, André Marette, Professor, Laval University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: MICA 2018-146
Record Dates: First submitted 2018-11-19; First posted 2018-11-27 (Actual); Last update posted 2020-03-30 (Actual); Status verified 2020-03

CONDITIONS: Overweight; Insulin Resistance; Microbiota; Endotoxemia; Metabolic Syndrome
MeSH Terms: conditions — Overweight; Insulin Resistance; Endotoxemia; Metabolic Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Cranberry (Experimental): Whole Cranberry Powder Supplements
  Interventions: Dietary Supplement: Cranberry powder
- Placebo (Placebo Comparator): Placebo
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Cranberry powder — 3 capsules /day of whole cranberry powder (500mg/each)
  Arms: Cranberry
Dietary Supplement: Placebo — 3 capsules/day of a placebo comparator
  Arms: Placebo

SUMMARY:
It is of major importance to refine prevention strategies in order to alleviate inflammation, insulin resistance and metabolic syndrome and it appear that improving gut health and microbiota represent a promising strategy. Cranberry-enriched diets may help prevent metabolic syndrome and its associated chronic diseases by a protective effect of gut health and microbiota. It is therefore highly relevant to test the hypothesis that a whole cranberry powder supplements (which include a mixture of polyphenols, free and fiber-associated proanthocyanidins, and fruits fibers) is associated with changes on the gut health and microbiota playing a major role in alleviating inflammation and obesity-associated metabolic disorders.

DETAILED DESCRIPTION:
Over the past decade it has become clear that the gut microbiota is a key determinant of obesity and that its perturbations by nutritional insults play a significant role in the development of metabolic complications such as insulin resistance, type 2 diabetes, cardiovascular diseases and non-alcoholic fatty liver disease. Indeed, there is growing amounts of studies that have shown that dysbiosis of the intestinal microbiota promotes obesity-linked chronic inflammation, and is causally related to diet-induced type 2 diabetes. Our group recently published that a polyphenol-rich cranberry extract exert striking effect on the gut microbiota of high-fat and high-sucrose fed mice, which was associated with prevention of diet-induced weight gain, visceral obesity, insulin resistance and hepatic steatosis. Notably, metagenomic analyses of feces of the cranberry extract-treated mice suggested that these metabolic effects were associated with a dramatic increase in the proportion of Akkermansia muciniphila, a dominant commensal bacterium in the intestinal mucus layer which has received particular attention in the last few years since its abundance is associated with improved metabolic health and beneficial responses to various interventions in both mice and humans with obesity and diabetes. Polyphenols are now recognized as potent molecules capable to protect against obesity-linked metabolic diseases and dysbiosis. Among polyphenols, there is increasing evidence supporting the beneficial impact of dietary proanthocyanidins. Cranberries being rich in proanthocyanidins, we believe that these phyto-elements could be associated to their beneficial effects. On the other hand, apart from the recognized beneficial effects of fibers on gut health, their association with high molecular proanthocyanidins could also contribute to their health benefits.

The main objective of this study is to investigate in a cross-over randomized placebo-controlled clinical trial the beneficial properties of a whole cranberry powder on gut microbiota, intestinal health and metabolic syndrome parameters in overweight men.

ELIGIBILITY:
Inclusion Criteria:

* overweight
* fasting insulin > 42 pmol/L
* non smoking
* Stable weight in the past 3 months

Exclusion Criteria:

* chronic diseases
* Taking drugs that could affect glucose or lipid metabolism
* Taking anti-inflammatory, immunosuppressant or anticoagulant drugs
* Inflammatory bowel disease
* vegetarians, vegan or following any restrictive dietary pattern or if they are big consumers of berries (>1 portion/day)
* taking pre- and probiotics
* antibiotics in the past 3 months or change in their regular medication
* Major surgery in the past 3 months
* taste aversion for cranberries or cranberry allergy or allergies to other ingredients used in the placebo

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2018-10-15 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
Change in Gut Microbiota Diversity | At the beginning and the end of each treatment (4 weeks each)
  Global variation of the fecal microbiota

SECONDARY OUTCOMES:
Change in Endotoxemia | At the beginning and the end of each treatment (4 weeks each)
  Plasma Lipopolysaccharides (LPS) and Lipopolysaccharide Binding Protein (LBP)
Change in Intestinal permeability | At the beginning and the end of each treatment (4 weeks each)
  Plasma zonulin
Change in Inflammation state of the tissue | At the beginning and the end of each treatment (4 weeks each)
  Fecal calprotectin and chromogranin
Change in Short chain fatty acids in the feces | At the beginning and the end of each treatment (4 weeks each)
  Measure short chain fatty acids in the feces
Change in Gut health and stool consistency | At the beginning and the end of each treatment (4 weeks each)
  Evaluation of gastrointestinal symptoms and stool consistency using standardized questionnaires
Change in Lipid profile | At the beginning and the end of each treatment (4 weeks each)
  Evaluation of plasma triglycerides (TG), Total cholesterol, LDL, HDL and Apolipoprotein B from the beginning to the end of two dietary treatment
Change in chronic inflammation | At the beginning and the end of each treatment (4 weeks each)
  Evaluation of plasma high sensitive C-Reactive Protein (hs-CRP)
Change in Glucose homeostasis | At the beginning and the end of each treatment (4 weeks each)
  Evaluation of plasma fasting glucose and insulin concentration

CONTACTS AND LOCATIONS:
Overall Officials: André Marette, Ph.D, Principal Investigator — Institute of nutrition and functional foods, Laval University
Locations (1):
- Institut sur la nutrition et les aliments fonctionnels, Québec, Canada